CLINICAL TRIAL: NCT01699503
Title: Indiana University Dementia Screening Trial: The IU CHOICE Study
Brief Title: Indiana University Dementia Screening Trial
Acronym: IU-CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nicole R. Fowler, PhD, Regenstrief Institute, IU Center for Aging Research Scientist, Regenstrief Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: R01AG040220-01A1 (NIH); 1R01AG040220-01A1 (NIH)
Record Dates: First submitted 2012-09-19; First posted 2012-10-03 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Dementia; Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Dementia; Alzheimer's Disease; Mild Cognitive Impairment; Screening
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Screening (No Intervention): Subjects who are randomized into the non-screening arm will receive the usual standard of care.
- Screening Group (Experimental): Subjects who are randomized into the screening arm of the study will be screened by the MIS. Subjects with MIS score of less than 5 points will be referred to the Collaborative Dementia Care Program for a subsequent diagnostic assessment, counseling and management.
  Interventions: Behavioral: Collaborative Dementia Care Program

INTERVENTIONS:
Behavioral: Collaborative Dementia Care Program — Much of the intervention, facilitated by care coordinator, is targeted to co-manage or support the practice behavior of primary care clinicians, enhance self-management skills of both the care-recipient and the informal caregiver, and maximize the coping behavior of the patient and the informal caregiver.
  Arms: Screening Group

SUMMARY:
The purpose of the study is to conduct a randomized clinical trial assessing the harms and benefits of screening for dementia, compared to no screening for dementia, among 4,000 older adults, cared for in typical, primary care practices.

DETAILED DESCRIPTION:
The objective of this proposal is to address the question of whether the benefits outweigh the harms of routine screening for dementia among older adults in primary care when the screening program is coupled with primary care practices prepared to provide care for those who screen positive.

The specific aim of the study is to conduct a pragmatic randomized clinical trial assessing the harms and benefits of screening for dementia, compared to no screening for dementia, among 4,000 typical, older adults, cared for in typical, primary care practices, prepared to deliver best practices dementia care.

Primary Specific Aim 1:

Test the impact of dementia screening on health-related quality of life of the patient at 12 months.

Primary Specific Aim 2:

Test the impact of dementia screening on the mood and anxiety symptoms of patient at 1 month (i.e., primary potential harms).

Secondary Aims: Estimate the cost effectiveness of dementia screening.

ELIGIBILITY:
Inclusion Criteria:

* adults age 65 and older;
* at least one office visit to their primary care physician within the previous year;
* no previous diagnosis of dementia or memory problem as determined by ICD-9 codes or the presence of prescription for anti-dementia medications (cholinesterase inhibitors or memantine);
* ability to consent to participate in the study; and
* ability to communicate in English

Exclusion Criteria:

* adults who are a permanent resident of a nursing facility;
* a serious mental illness such as bipolar disorder or schizophrenia as determined by the presence of related ICD-9 codes indicative of such an illness; or
* a pre-existing diagnosis of dementia or cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4005 (Actual)
Dates: Start 2012-10; Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, MPH, Principal Investigator — Regenstrief Institute, Inc.
Locations (3):
- United States (3):
  - IU Health-Primary Care Clinics, Indianapolis, Indiana
  - Wishard Health Services-Primary Care Clinics, Indianapolis, Indiana
  - IU Health Arnett Primary Care Clinics, West Lafayette, Indiana

REFERENCES:
- [Background] Boustani M, Perkins AJ, Monahan P, Fox C, Watson L, Hopkins J, Fultz B, Hui S, Unverzagt FW, Callahan CM, Hendrie HC. Measuring primary care patients' attitudes about dementia screening. Int J Geriatr Psychiatry. 2008 Aug;23(8):812-20. doi: 10.1002/gps.1983. PMID 18232061
- [Background] Boustani M, Peterson B, Hanson L, Harris R, Lohr KN; U.S. Preventive Services Task Force. Screening for dementia in primary care: a summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Jun 3;138(11):927-37. doi: 10.7326/0003-4819-138-11-200306030-00015. PMID 12779304
- [Background] Boustani MA, Justiss MD, Frame A, Austrom MG, Perkins AJ, Cai X, Sachs GA, Torke AM, Monahan P, Hendrie HC. Caregiver and noncaregiver attitudes toward dementia screening. J Am Geriatr Soc. 2011 Apr;59(4):681-6. doi: 10.1111/j.1532-5415.2011.03327.x. Epub 2011 Mar 25. PMID 21438862
- [Background] Fowler NR, Boustani MA, Frame A, Perkins AJ, Monahan P, Gao S, Sachs GA, Hendrie HC. Effect of patient perceptions on dementia screening in primary care. J Am Geriatr Soc. 2012 Jun;60(6):1037-43. doi: 10.1111/j.1532-5415.2012.03991.x. PMID 22690979
- [Derived] Fowler NR, Perkins AJ, Gao S, Sachs GA, Boustani MA. Risks and Benefits of Screening for Dementia in Primary Care: The Indiana University Cognitive Health Outcomes Investigation of the Comparative Effectiveness of Dementia Screening (IU CHOICE)Trial. J Am Geriatr Soc. 2020 Mar;68(3):535-543. doi: 10.1111/jgs.16247. Epub 2019 Dec 2. PMID 31792940
- [Derived] Fowler NR, Harrawood A, Frame A, Perkins AJ, Gao S, Callahan CM, Sachs GA, French DD, Boustani MA. The Indiana University Cognitive Health Outcomes Investigation of the Comparative Effectiveness of dementia screening (CHOICE) study: study protocol for a randomized controlled trial. Trials. 2014 Jun 6;15:209. doi: 10.1186/1745-6215-15-209. PMID 24903469

RESULTS

PARTICIPANT FLOW:
Groups:
- Screening Group: Subjects who are randomized into the screening arm of the study will be screened by the Memory Impairment Screen (MIS). Subjects with MIS score of less than 5 points will be referred to the Collaborative Dementia Care Program for a subsequent diagnostic assessment, counseling and management.
  Collaborative Dementia Care Program: Much of the intervention, facilitated by care coordinator, is targeted to co-manage or support the practice behavior of primary care clinicians, enhance self-management skills of both the care-recipient and the informal caregiver, and maximize the coping behavior of the patient and the informal caregiver.
Period: Overall Study
Arm/Group | Screening Group | No Screening
Started | 2008 | 1997
Baseline | 1723 | 1693
1 Month Follow-up | 998 | 1022
6 Month Follow-up | 903 | 893
Completed | 1008 | 992
Not Completed | 1000 | 1005
Not completed — Death | 31 | 40
Not completed — Withdrawal by Subject | 65 | 57
Not completed — Lost to Follow-up | 121 | 117
Not completed — Excluded due to quality | 783 | 791

BASELINE CHARACTERISTICS:
Groups:
- Screening Group: Subjects who are randomized into the screening arm of the study will be screened by the Memory Impairment Screen(MIS). Subjects with MIS score of less than 5 points will be referred to the Collaborative Dementia Care Program for a subsequent diagnostic assessment, counseling and management.
  Collaborative Dementia Care Program: Much of the intervention, facilitated by care coordinator, is targeted to co-manage or support the practice behavior of primary care clinicians, enhance self-management skills of both the care-recipient and the informal caregiver, and maximize the coping behavior of the patient and the informal caregiver.
- Total: Total of all reporting groups
Arm/Group | Screening Group | No Screening | Total
Number analyzed (Participants) | 1723 | 1693 | 3416
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (7.0) | 74.1 (6.8) | 74.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1167 | 1089 | 2256
  Male | 556 | 604 | 1160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 526 | 530 | 1056
  White | 1164 | 1137 | 2301
  Other | 31 | 24 | 55
  Missing | 2 | 2 | 4
Co-morbidity status, no (%) [Count of Participants; unit: Participants]
  Cancer | 379 | 392 | 771
  Chronic Lung Disease/Emphysema/COPD | 698 | 655 | 1353
  Congestive Heart Failure | 301 | 311 | 612
  Peripheral Vascular Disease | 253 | 257 | 510
  Coronary Artery Disease | 567 | 585 | 1152
  Diabetes | 731 | 685 | 1416
  Hypertension | 1428 | 1383 | 2811
  Stroke | 390 | 393 | 783
Charlson co-morbidity score, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — The Charlson Comorbidity Index is a method of predicting mortality by classifying or weighting co-morbid conditions. Each of the 12 comorbidity categories has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. Scores range from 0-24. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
  units on a scale | 2.7 (2.8) | 2.8 (3.0) | 2.8 (2.9)
Education level, no (%) [Count of Participants; unit: Participants] — Population: 22 participants refused to answer their education level
  Participants
    number analyzed (Participants) | 1712 | 1682 | 3394
    Less than high school | 363 | 357 | 720
    High school | 571 | 556 | 1127
    Some college or college degree | 778 | 769 | 1547
Self-reported social support¥, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — Measured with the MOS-5 Social Support Inventory. The MOS Social Support Survey, a brief multidimensional self administered instrument, was selected to assess perceived support.The higher the score, the more perceived support. Scores range from 0-100.
  Compute raw score by adding scores on these 5 items Raw scores on this scale range from 5-25. Compute transformed score as follows: [(Raw score-5)/20] x 100
  units on a scale | 21.0 (4.5) | 20.8 (4.6) | 20.9 (4.6)
Study Site, no (%) [Count of Participants; unit: Participants]
  Urban, safety net health system | 725 | 709 | 1434
  Rural health system | 653 | 624 | 1277
  Suburban and urban academic health system | 345 | 360 | 705
Health-related quality of life, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — Measured by the Health Utilities Index (HUI). A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death.The HUI classification system is comprised of 8 attributes - Vision, Hearing, Speech, Ambulation, Dexterity, Emotion, Cognition and Pain - each with 5 or 6 levels of ability/disability.Single-attribute scores of morbidity are defined on a scale such the worst level has a score of 0.00 and the best level has a score of 1.00. The higher the score, the better the health related quality of life.
  units on a scale | 0.67 (0.27) | 0.67 (0.27) | 0.67 (0.27)
Depressive symptoms, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — Measured by the Patient Health Questionaire-9 (PHQ-9). The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).Scores range from 0-27. A higher score means higher depressive symptoms.
  units on a scale | 3.23 (4.07) | 3.06 (3.69) | 3.15 (3.89)
Anxiety, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — Measured by the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is a valid and efficient tool for screening for Generalized Anxiety Disorder and assessing its severity in clinical practice and research.Scores range from 0-21, with 0-3 points for each of seven questions. A higher score is associated with more severe anxiety.
  units on a scale | 1.79 (3.33) | 1.77 (3.19) | 1.78 (3.26)

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life (HRQOL)
Description: The primary outcome measure will be the HRQOL measured at baseline, 1, 6 and 12 months among the entire 4,000 enrollees. The study will use the 15-item Health Utility Index (HUI) to determine the subject's HRQOL. The HUI is a generic, utility-based HRQOL instrument applied in patients with a wide range of medical conditions. It has eight attributes: Vision, hearing, speech, ambulation, dexterity, emotion, cognition and pain. The individual health domain scores range from 0.00 (maximum impairment) to 1.00 (no impairment) and the multi-attribute (HUI index) scores, a multiplicative function of individual attribute levels, range from 0.36 to 1.00 with anchors 0.00 = dead and 1.00 = perfect health.
Time Frame: 1 month, 6 months, 12 months
Population: The number analyzed for each row excludes those participants who died, withdrew, were lost to follow-up, or were excluded due to quality at each time point in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Screening Group | No Screening
Number analyzed (Participants) | 1723 | 1693
units on a scale
  1 Month: number analyzed (Participants) | 974 | 1000
  1 Month | 0.71 (0.24) | 0.69 (0.26)
  6 Month: number analyzed (Participants) | 885 | 875
  6 Month | 0.69 (0.26) | 0.70 (0.25)
  12 Month: number analyzed (Participants) | 993 | 976
  12 Month | 0.67 (0.27) | 0.68 (0.26)

2. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a nine-item depression scale with a total score from 0 to 27. It has a good internal consistency and test-retest reliability; as well as convergent, construct, criterion, procedural and factorial validity for the diagnosis of major depression. A higher score is associated with more severe depression.
Time Frame: 1 month, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Screening Group | No Screening
Number analyzed (Participants) | 1723 | 1693
units on a scale
  1 Month: number analyzed (Participants) | 996 | 1022
  1 Month | 2.33 (3.22) | 2.46 (3.27)
  6 Month: number analyzed (Participants) | 903 | 893
  6 Month | 2.50 (3.43) | 2.45 (3.34)
  12 Month: number analyzed (Participants) | 1006 | 992
  12 Month | 2.74 (3.69) | 2.82 (3.71)

3. Primary Outcome: Generalized Anxiety Disorder Scale (GAD-7)
Description: The GAD-7 is a seven-item anxiety scale with a total score from 0 to 21. It has a good internal consistency and test-retest reliability; as well as convergent, construct, criterion, procedural and factorial validity for the diagnosis of general anxiety disorder. A higher score is associated with more severe anxiety.
Time Frame: 1 month, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Screening Group | No Screening
Number analyzed (Participants) | 1723 | 1693
units on a scale
  1 Month: number analyzed (Participants) | 997 | 1022
  1 Month | 1.16 (2.57) | 1.24 (2.54)
  6 Month: number analyzed (Participants) | 903 | 893
  6 Month | 1.24 (2.60) | 1.13 (2.37)
  12 Month: number analyzed (Participants) | 1005 | 992
  12 Month | 1.31 (2.77) | 1.45 (2.83)

4. Secondary Outcome: Number of Participants With Health Care Utilization
Description: The study team will obtain consent at enrollment from all subjects for permission to review their medical records. The Indiana Network for Patient Care (a fully operational Health Information Exchange) will also be used to identify any episode of ambulatory or acute care that occurred within the following 12 months of enrollment date.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Group | No Screening
Number analyzed (Participants) | 1723 | 1693
Participants
  Patients with at least 1 ED visit in 12 months | 510 | 512
  Patients with at least 1 hospitalization in 12 mo | 336 | 333

5. Secondary Outcome: Number of Participants With an Advance Directive at 12 Months
Description: The study team will measure the subjects' advanced care planning including having power attorney for health care and/or financial affairs, having a living will, and having life and additional insurance policies at 12 months.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Group | No Screening
Number analyzed (Participants) | 992 | 1008
Participants | 653 | 644

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Screening Group | No Screening
All-Cause Mortality (participants affected / at risk) | 21/1723 | 25/1693
Serious Adverse Events (participants affected / at risk) | 52/1723 | 47/1693
Other Adverse Events (participants affected / at risk) | 0/1723 | 0/1693
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening Group (N=1723) | No Screening (N=1693)
Incident Severe Depression ( (Psychiatric disorders) | 34 | 28 — Severe Depression is defined as PHQ-9 score of 15+
Incident Severe Anxiety (Psychiatric disorders) | 18 | 19 — Severe Anxiety is defined as GAD-7 score of 15 - 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT01699503/Prot_SAP_000.pdf